CLINICAL TRIAL: NCT06201819
Title: Liraglutide Effectiveness in Preoperative Weight-loss for Patients With Severe Obesity Undergoing Bariatric-metabolic Surgery.
Brief Title: Liraglutide Effectiveness in Preoperative Weight-loss for Bariatric-metabolic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unidad de Cirugia Bariatrica Hospital Civil Dr. Juan I. Menchaca (Other)
Responsible Party: Principal Investigator, Jose Daniel Reyes Blandón, Bariatric Surgery Resident, Unidad de Cirugia Bariatrica Hospital Civil Dr. Juan I. Menchaca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI-008-20161212
Record Dates: First submitted 2023-12-14; First posted 2024-01-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss; Bariatric Surgery Candidate; Obesity, Morbid
Keywords: Preoperative weight loss
MeSH Terms: conditions — Weight Loss; Obesity, Morbid | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: quasi-experimental prospective before-and-after study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with morbid obesity in bariatric surgery preparation protocol (Experimental): All patients with body mass index >48 kg/m2 in preoperative protocol for bariatric surgery using liraglutide for preoperative weight loss
  Interventions: Drug: Liraglutide injection

INTERVENTIONS:
Drug: Liraglutide injection — Liraglutide (GLP-1 analog) injection during 3 months

SUMMARY:
Severe obesity is associated with considerable reduction of wellbeing and life expectancy. People living with severe obesity tend to die 8 to 10 years earlier. Preoperative management of patients living with severe obesity can be challenging and proper weight-loss may help obtain better outcomes and less morbidity. The effectiveness of GLP-1 analogue Liraglutide in preoperative weight-loss was evaluated in the study.

DETAILED DESCRIPTION:
Objective:

Determine liraglutide effectiveness for preoperative weight-loss in patients with severe obesity undergoing bariatric-metabolic surgery.

Methods:

It is a single center, quasi-experimental prospective before-and-after study. All patients were assigned the same pharmacological treatment with liraglutide, initiating dosing with 0.6 mg per day escalating 0.6 mg every week up to 3.0 mg. The treatment dose was delivered once daily via subcutaneous injection for 3 months (12 weeks). Weight-loss and percentage weight-loss was evaluated monthly using bioelectric impedance (BIA) final result at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI greater than 48 kg/m2 in pre-surgical protocol for bariatric surgery of the Bariatric and Metabolic Surgery Unit of the Civil Hospital of Guadalajara "Dr. Juan I. Menchaca

Exclusion Criteria:

* Patients under 18 years of age or over 65 years of age.

  * Pregnant patients.
  * Patients who do not agree to give their consent and take part in the study.
  * Patients with allergy to liraglutide, multiple endocrine neoplasia type 2 and medullary thyroid cancer, gallstones.

Removal:

* Patients who decide to abandon the study.
* Patients who do not follow the instructions or do not adhere to the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Preoperative weight changes | 3 months
  Total body weight change during the drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Cirugia Bariatrica y Metabolica del Hsopital Civil Dr. Juan I. Menchaca, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol
Time Frame: 3 months
Access Criteria: Available on request to the main author